CLINICAL TRIAL: NCT05720000
Title: Effect of Photobiomodulation Associated With Polydioxanone Thread in the Treatment of Glabellar Wrinkles: Clinical, Randomized, Controled, Double Blind Trial
Brief Title: Use of Red Light Emitting Diode (LED) and Polydioxanone Thread in Glabellar Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Christiane Pavani, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCG
Record Dates: First submitted 2022-12-24; First posted 2023-02-09 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Skin Wrinkling; Edema
Keywords: polydioxanone thread; LED; photobiomodulation (PBM); Glabellar line
MeSH Terms: conditions — Edema | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: All participants will receive PDO thread at glabella. Immediately after application, the participants will receive the intervention related to their treatment group, according to the allocation given by randomization. After randomization, the study population will be divided into two groups (n=20 per group), which are: (1) Group A - PDO thread + PBM with red LED, (2) PDO thread + PBM sham. The treatment will be performed twice a week for 30 days, in total 9 sessions.
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the participants involved in the study, nor the outcomes assessor will be aware of the groups formed, as well as the treatments received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDO thread with active red LED photobiomodulation (PBM) (Experimental): Participants will receive the PDO thread and the intervention with PBM using red light (Newskin, MMO) 150 mW, 2J per point, 4J/cm2, 10 points, twice a week.
  Interventions: Device: Photobiomodulation; Procedure: PDO thread
- PDO thread with sham photobiomodulation (PBM) (Sham Comparator): Participants will receive the PDO thread and the simulated intervention with PBM using Newskin, MMO.
  Interventions: Procedure: PDO thread

INTERVENTIONS:
Device: Photobiomodulation — Patient will receive the application of the low-power 660 nm Newskin MMO red LED in the immediate postoperative period. The application will be made punctually over the entire length of the wire, which measures 5 cm, totaling 10 application points with 1 cm of distance between them. The LED application will be repeated twice a week, with a minimum interval of 48 hours, totaling 9 laser applications over 30 days.
  Arms: PDO thread with active red LED photobiomodulation (PBM)
Procedure: PDO thread — The participant's face will be cleaned with a 0.2% chlorhexidine solution. 0.1 ml of injectable anesthetic (2% lidocaine hydrochloride without vasoconstrictor, XYlestesin) will be administered in the skin layer at the point of incision in the glabellar region with a 30-gauge needle. A subincision will be made with a 21-gauge cannula in the glabellar ridge and then an injectable thread will be applied in the deep dermal layer below the glabellar ridge in the same direction as it.

SUMMARY:
Physical appearance is a factor that contributes to an individual's self-esteem. Maintaining a healthy appearance is a growing quest by the population, and aging is the main cause of discomfort for men and women. There are several aesthetic treatments capable of mitigating or delaying the effects of aging in all its layers of alteration (dermis, hypodermis, musculature and bone), and the combination of therapies has been increasingly proposed in search of a positive synergy. The dermal application of polydioxanone threads (PDO) and the low-power red LED (photobiomodulation - PBM) are individual options of resources for which there already are reports in the literature about their mechanisms of action in the proliferation of fibroblasts and collagen production. However, the joint application of these techniques requires further studies.

A total of 40 patients, aged between 30 and 60 years old, phototypes I-IV in Fitzpatrick scale, Glogau 3-4, presenting static wrinkle at the glabellar region will be recruited and distributed among 2 groups: PDO thread + PBM or PDO thread + sham PBM. The treatments will consist of 30 days, with one application of PDO thread and PBM twice a week (total of 9 sessions).

DETAILED DESCRIPTION:
This is a controled, randomized, double blind, two arms clinical trial. The main objective of this study is to evaluate the effect of PBM with red light associated to PDO threads in individuals with static wrinkles in the glabellar region in terms of oedema, dermal thickening and PDO thread hydrolysis.

The sample will be divided into 2 groups: Group 1 will receive PDO thread and PBM with Red LED (Newskin, MMO), 150 milliwatt (mW), 2 Joule (J) per point, 4 J/cm² , 10 points per session, Group 2 will receive PDO thread and PBM sham. A total of 40 patients with glabellar wrinkle, aged 30 to 60 will be included. The treatments will consist of 9 sessions, twice a week for 30 days. The oedema and dermal thickness will be evaluated by linear ultrasound (10-14 MegaHertz (MHz), Mobisson). Photographic records will also be made.

ELIGIBILITY:
Inclusion Criteria:

* both genders
* aged between 30 and 60 years,
* Fitzpatrick skin phototype I - IV,
* levels 3 and 4 in the aging classification according to Glogau,
* presenting glabellar static wrinkles (permanent wrinkles)
* who do not have uncompensated comorbidities.

Exclusion Criteria:

* decompensated diabetes, lupus, HIV positive, hepatitis, high blood pressure, neurological disorders, active neoplasms,
* tendency to develop keloids,
* menopause, pregnant women,
* participants who have absorbable threads (applied less than 3 months ago) or definitive at glabella,
* who have PMMA (polymethylmethacrylate) application in any region of the face,
* who are undergoing treatment with any type of laser therapy in any areas of the body,
* participants who are undergoing aesthetic or dermatological treatment on the face,
* participants who are using anti-inflammatories and corticoids in a window of 30 days before and after the procedure,
* participants using isotretinoin in the last 6 months.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Edema assessed by Ultrasound | Before treatment (day 0)
  Ultrasound transversal measurement from epidermis to the beginning of muscle tissue.
Edema assessed by Ultrasound | 24 hours after PDO thread application (day 1)
  Ultrasound transversal measurement from epidermis to the beginning of muscle tissue.

SECONDARY OUTCOMES:
dermis thickness | Before treatment (day 0)
  Ultrasound transversal measurement from epidermis to the beginning of muscle tissue.
dermis thickness | day 90
  Ultrasound transversal measurement from epidermis to the beginning of muscle tissue.
PDO thread hydrolysis | day 180
  Ultrasound identification of presence or absence of the thread
Photos | Before treatment (day 0)
  Image registration of the region treated
Photos | 24 hours after PDO thread application (day 1)
  Image registration of the region treated
Photos | day 90
  Image registration of the region treated
Photos | day 180
  Image registration of the region treated

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Pavani, PhD, Study Director — University of Nove de Julho
Locations (1):
- Clinic Cursos, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices will be shared). The sharing will begin 3 months following article publication. Researchers who provide a methodologically sound proposal will have the access. Proposals should be directed to chrispavani@gmail.com. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The sharing will begin 3 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.